CLINICAL TRIAL: NCT03563664
Title: Effect of Danazol on Endometrial αvβ3 Integrin Expression in Patients With Unexplained Recurrent Implantation Failure - A Self-controlled Clinical Trial
Brief Title: Effect of Danazol on Endometrial αvβ3 Integrin Expression in Patients With Unexplained Recurrent Implantation Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohammed mahmoud samy, Lecturer in Obstetrics and Gynecology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIF-Danazol
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Unexplained Infertility
MeSH Terms: interventions — Danazol

STUDY DESIGN:
Intervention Model Description: 38 ovulatory patients with unexplained recurrent implantation failure were recruited. Endometrial αvβ3 integrin expression (using immunohistochemically stained endometrial biopsy) was compared before and after treatment with danazol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): 38 ovulatory patients with unexplained recurrent implantation failure were recruited. Pre-treatment endometrial biopsy and immunohistochemical examination for endometrial αvβ3 integrin expression (using immunohistochemically stained endometrial biopsy) was done. After treatment with danazol (Danol® 200mg capsules, Sanofi, Guildford, UK) in daily dosage of 400 mg for 12 weeks, post-treatment endometrial biopsy and immunohistochemical examination was repeated and compared with previous results.
  Interventions: Procedure: Pre-treatment endometrial biopsy; Drug: Danazol; Procedure: Post-treatment endometrial biopsy

INTERVENTIONS:
Procedure: Pre-treatment endometrial biopsy — Timed suction endometrial biopsy was obtained from participants via Wallach Endocell® 908014A endometrial cell sampler timed during the implantation window of the pretreatment cycle; followed by immunohistochemical staining using immunoperoxidase staining incorporating avidin-biotin complex (ABC) method.
Drug: Danazol — Participants were treated with danazol (Danol® 200mg capsules, Sanofi, Guildford, UK) in daily dosage of 400 mg for 12 weeks.
Procedure: Post-treatment endometrial biopsy — Post-treatment suction endometrial biopsy was obtained during the implantation window following the first ovulation after danazol treatment, timed, processed and stained as described previously.

SUMMARY:
This study investigates the presence of a possible link between treatment with danazol and expression of endometrial αvβ3 integrin which might allow tailoring of danazol treatment to the subset of repeated IVF/ET failure that might benefit most from it.

38 eligible ovulatory women were recruited aged 20 - 38 years with unexplained recurrent implantation failure (RIF). Timed suction endometrial biopsy was obtained from participants during the implantation window of the pretreatment cycle, followed by immunohistochemical staining for endometrial αvβ3 integrin expression, scored using H-score.

Participants were treated with danazol (Danol® 200mg capsules, Sanofi, Guildford, UK) in daily dosage of 400 mg for 12 weeks. Post-treatment suction endometrial biopsy was obtained during the implantation window following the first ovulation after danazol treatment and endometrial αvβ3 integrin expression was compared to the pretreatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-38 yrs
* Unexplained recurrent implantation failure (RIF), defined as failure to achieve an intrauterine gestational sac recognized by ultrasonography after transfer of at least four good-quality embryos (defined as those with four or five blastomeres on day 2, seven or more cells on day 3, ≤ 20% anucleated fragments and absence multinucleated blastomeres) in a minimum of three fresh or frozen IVF cycles after exclusion of other causes of RIF (as depicted by normal transvaginal ultrasonography, hysteroscopy, hysterosalpingography, laparoscopic findings, male and female karyotypic examination, endocrinological profile during ovarian stimulation and negative anti-cardiolipin antibody IgM/IgG, lupus anticoagulant, thrombophilia screening (including protein C, protein S, anti thrombin III and factor V leiden) and normal male semen analysis as depicted by 2010 WHO criteria for semen analysis and sperm DNA fragmentation testing).

Exclusion Criteria:

* Anovulation
* Contraindications to treatment with danazol (including chronic liver disease, congestive heart failure, dyslipidemia or history/current thrombo-embolic disease)
* Medical comorbidities (e.g. autoimmune disorders, diabetes mellitus, etc)
* Patients who underwent induction of ovulation / received hormonal treatment during the previous three months

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
H-score | 12 weeks
  Stained sections were evaluated by the same pathologist for the intensity of brownish cytoplasmic and membranous staining of the endometrial components using the semi-quantitative scoring system originally described by Budwit-Novotny et al., H-score [6], calculated using the formula H-score=∑▒〖P_i (i+1)〗 where i is the staining intensity valued as 0, absent; 1+, weak, but detectable above control; 2+, moderate and 3+, strong; and Pi is the percentage of epithelial cells stained with each intensity (varying from 0 to 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy, MD, Principal Investigator — M Samy
Locations (1):
- Ain SHams Maternity Hospital, Cairo, Abbaseya, Egypt